CLINICAL TRIAL: NCT04759703
Title: Treatment of Restless Legs Symptoms With Pramipexole to Improve the Outcomes of Protracted Opioid Withdrawal in OUD: A Pilot Double-blind, Randomized Clinical Trial
Brief Title: Treatment of Restless Legs Symptoms With Pramipexole to Improve the Outcomes of Protracted Opioid Withdrawal in OUD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: An interim analysis indicated that we would need to enroll more subjects than our initial enrollment target, in order to demonstrate a significant treatment effect. Due to these results, we have decided to terminate this protocol.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Winkelman, MD, PhD, Chief, Sleep Disorders Clinical Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P002928; R21DA052861 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorder; Restless Legs Syndrome; Opioid-use Disorder; Opioid Withdrawal
Keywords: Pramipexole
MeSH Terms: conditions — Sleep Wake Disorders; Restless Legs Syndrome; Opioid-Related Disorders | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pramipexole (Experimental): Medication arm; 0.25 of pramipexole
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Placebo arm; 0.25 mg of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole — 0.25 mg pramipexole tablets
  Other Names: Mirapex
  Arms: Pramipexole
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
The investigators propose to test the use of pramipexole in patients being treated for Opioid Use Disorder to test its ability to reduce symptoms of both Restless Legs Syndrome and protracted opioid withdrawal and thereby promote initiation, engagement, and retention in treatment.

DETAILED DESCRIPTION:
This is a parallel, two-arm, double-blind, randomized placebo-controlled 2-week trial investigating the effects of pramipexole 0.25-0.5 mg on Restless Legs Syndrome (RLS) symptoms in patients suffering from opioid withdrawal. The investigators hypothesize that pramipexole is an effective treatment for RLS symptoms in Opioid Use Disorder (OUD) patients during post-detox clinical stabilization. Further, the investigators hypothesize that treatment of RLS in this context will also improve overall symptoms of opioid withdrawal.

RLS is a sensory-motor neurological disorder characterized by an irresistible urge to move the legs. The investigators have recently confirmed anecdotal reports that RLS is common among patients with OUD experiencing opioid withdrawal. Dopamine agonists such as pramipexole are efficacious and first-line FDA-approved treatments in low doses for RLS.

Recruitment and enrollment will occur at the Gavin Foundation Clinical Stabilization Services (CSS) in Quincy, Massachusetts. Eligible patients will be randomized to two weeks of pramipexole or placebo after an initial 3-day screening period and will be asked to complete 5 remote study visits over video or phone. Participants will be asked to complete sleep diaries and questionnaires at various points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of any ethnic origin.
2. Written informed consent is obtained
3. Speaks and writes in English
4. A willingness and ability to comply with study procedures.
5. Age 18-75 years
6. Patients with diagnosed OUD who have undergone primary detoxification for their OUD in the Gavin Acute Treatment Service (ATS), have been transferred to the Gavin Clinical Stabilization Service (CSS), and have some persistent opioid withdrawal as indicated by a Subjective Opiate Withdrawal Scale (SOWS) >1 on Day 1
7. Diagnosis of RLS from the Hening Telephone Diagnostic Interview (HTDI) with subsequent confirmation by clinical interview conducted by a study physician
8. International Restless Legs Syndrome Severity Scale (IRLS) Symptoms subscale score of >15 for three consecutive days prior to randomization

Exclusion Criteria:

1. Receiving opioid-agonist medications at transfer to the CSS
2. Pregnant
3. Participants with active or unstable major psychiatric disorder other than OUD, who, in the investigators' judgment, require further treatment
4. Use of dopaminergic agonists or antagonists within the last 30 days
5. Alcohol use disorder within the last 30 days
6. History of being treated for RLS, specifically with dopamine agonist medications
7. Methamphetamine or benzodiazepine dependence in the last 30 days
8. Neurological disorder or cardiovascular disease raising safety concerns about use of pramipexole and/or judged to interfere with ability to assess efficacy of the treatment
9. Medical instability considered to interfere with study procedures
10. Stage 3, 4, or 5 renal insufficiency
11. Participation in this study on a previous admission to the CSS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD/PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Gavin Foundation Clinical Stabilization Services, Quincy, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make data available on a public database. Outside investigators should submit their request in writing to the PI. A data-sharing agreement will be required. The request must be in accordance with Mass General Brigham (MGB) Policies and Harvard Medical School (HMS) Guidelines. Such datasets will not contain identifying information per the regulations outlined in HIPPA, and permission will be obtained from study participants to share their data with researchers outside MGB. Per standard MGB policies, the investigators will require a data-sharing agreement from any investigator or entity requesting the data; this agreement will include: (i) a commitment to using the data only for research purposes and not to identify any individual participant; (ii) a commitment to securing the data using appropriate computer technology; and (iii) a commitment to destroying or returning the data after analyses are completed.
Time Frame: Per the NIH Policy on Data Sharing, the investigators will make the datasets available to other investigators following publication of the final study results.
Access Criteria: Requests must be in accordance with Mass General Brigham Policies and Harvard Medical School Guidelines.

REFERENCES:
- [Background] Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse. 1987;13(3):293-308. doi: 10.3109/00952998709001515. PMID 3687892
- [Background] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342
- [Background] Hening WA, Allen RP, Washburn M, Lesage S, Earley CJ. Validation of the Hopkins telephone diagnostic interview for restless legs syndrome. Sleep Med. 2008 Mar;9(3):283-9. doi: 10.1016/j.sleep.2007.04.021. Epub 2007 Jul 17. PMID 17644424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Gavin Foundation Clinical Stabilization Services in Quincy. A total of 175 patients were referred, 93 were screened, and 75 patients enrolled.
Pre-assignment Details: After screening, 18 of the 93 patients were found ineligible and 35 withdrew or failed. 40 completed post randomization baseline data.
Period: Overall Study
Arm/Group | Pramipexole | Placebo
Started | 20 | 20
Completed | 13 | 11
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Of 75 enrolled, 35 participants Withdrew/Failed before baseline data collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years at screening date
  Years | 39.1 (9.6) | 35.2 (5.8) | 37.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 13 | 17 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 15 | 17 | 32
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 20 | 40
Subjective Opiate Withdrawal Scale (SOWS) [Mean (Standard Deviation); unit: scores on a scale] — Subjective Opiate Withdrawal Scale (SOWS)
  Self-administered scale for grading opioid withdrawal symptoms. Scored from 0-64. Summed from 16 sub-scale questions from 0 to 4.
  Mild Withdrawal = score of 1 - 10 Moderate withdrawal = 11 - 20 Severe withdrawal = 21 - 30+
  scores on a scale | 21.18 (10.00) | 26.40 (10.61) | 23.93 (10.52)
International Restless Legs Syndrome Study Group Rating Scale (IRLS) [Mean (Standard Deviation); unit: scores on a scale] — Subjective assessment of primary features of restless legs syndrome, intensity and frequency, associated sleep problems
  Scored form 0-40. Summed from 10 sub-scale questions rated by the patient from 0 to 4.
  Very severe=31-40 points Severe=21-30 points Moderate=11-20 points Mild=1-10 points None=0 points
  scores on a scale | 14.94 (1.99) | 14.71 (1.89) | 14.85 (1.92)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline Subjective Opiate Withdrawal Scale (SOWS) at 2 Weeks
Description: The Subjective Opiate Withdrawal Scale (SOWS) is a 16-item self-administered instrument.
  Self-administered scale for grading opioid withdrawal symptoms. Scored from 0-64. Summed from 16 sub-scale questions rated by the patient from 0 to 4.
  Mild Withdrawal = score of 1 - 10 Moderate withdrawal = 11 - 20 Severe withdrawal = 21 - 30+
  Change in SOWS score (2 weeks minus baseline)
Time Frame: baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pramipexole: Medication arm; 0.25mg of pramipexole
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 13 | 11
scores on a scale | -11.60 (11.88) | -18.28 (13.41)

2. Primary Outcome: Change From Baseline International RLS Severity Score (IRLS) at 2 Weeks
Description: The International Restless Legs Syndrome Study Group Rating Scale (IRLS) is a 10-item patient-reported questionnaire designed to assess the severity of restless legs syndrome symptoms. Each item is scored from 0 (no symptoms) to 4 (very severe), for a total score range of 0 to 40, with higher scores indicating greater symptom severity. A negative change from baseline represents symptom improvement.
  Very severe=31-40 points Severe=21-30 points Moderate=11-20 points Mild=1-10 points None=0 points
  Change 2 weeks IRLS score minus baseline IRLS score
Time Frame: baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 13 | 11
scores on a scale | -7.04 (3.44) | -9.15 (6.56)

ADVERSE EVENTS:
Time Frame: From enrollment through study termination, up to 2 weeks after randomization
Description: Adverse events were collected daily by systemic assessment during inpatient stay and study visits.
Arm/Group | Pramipexole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 15/20 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=20) | Placebo (N=20)
Stomach cramps (Gastrointestinal disorders) | 4 | 3 — Self-reported, mild to moderate
Constipation (Gastrointestinal disorders) | 2 | 0 — Self-reported, mild
Nausea (Gastrointestinal disorders) | 4 | 1
Headaches (Nervous system disorders) | 2 | 1
Worsened RLS (Nervous system disorders) | 1 | 0
Drowsiness (General disorders) | 3 | 1
Jumpiness (Nervous system disorders) | 0 | 1
Muscle twitches (Nervous system disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Vivid Dreams (Psychiatric disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early and did not complete planned enrollment. There was a target enrollment of 160, but the study only got to 75 enrolled. Of those 75, only 40 received treatment (20 pramipexole, 20 placebo). Limited sample size limits reliability of analyses and adverse events may not be representative of the broader study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT04759703/Prot_SAP_000.pdf